CLINICAL TRIAL: NCT02735993
Title: Cardiac REgistry of Celution Device for the Processing of Adipose-derived Regenerative Cells: Treatment and Evaluation (CREATE)
Brief Title: Cardiac REgistry of Celution Device for the Processing of Adipose-derived Regenerative Cells
Acronym: CREATE
Status: Withdrawn | Type: Observational
Why Stopped: Corporate decision
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: CREATE
Record Dates: First submitted 2016-03-15; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Heart Failure; Coronary Artery Disease
Keywords: Celution; ADRC; Heart Failure; Device
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

SUMMARY:
This cardiac registry study will collect information from patients with ischemic or non-ischemic heart failure that have been treated with adipose-derived regenerative cells (ADRCs) delivered via intramyocardial injection.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 20 and < 80 years of age
* Significant multi-vessel coronary artery disease not amenable to percutaneous or surgical revascularization OR idiopathic dilated cardiomyopathy
* Symptoms of heart failure (e.g. NYHA Stages of Heart Failure Class II or III)
* On maximal medical therapy for heart failure and if present, anginal symptoms
* Hemodynamic stability (SBP ≥ 90 mm/Hg, HR <110 beats/min)
* Ejection fraction ≤ 45%
* Left ventricular wall thickness > 5 mm at the target site(s) for cell injection, confirmed by Contrast Echo within 4 weeks prior to enrollment, and free of thrombus

Exclusion Criteria:

* Vascular anatomy and/or peripheral artery disease that prevents or impedes cardiac catheterization
* Aortic or mitral valve disease where valve replacement is indicated
* Presence of mechanical aortic or mitral valves
* Presence of aortic dissection
* Planned staged treatment of CAD or other therapeutic intervention on the heart within the subsequent 3 months
* TIA or stroke within 30 days prior to the procedure
* ICD placement or ablation therapy within 30 days prior to the procedure
* Acute coronary syndrome (ACS) or a myocardial infarction in the 30 days prior to the procedure
* Revascularization within 30 days prior to intramyocardial injection of ADRCs
* Pregnant or lactating status. Pregnancy as determined by a positive pregnancy test at screening or baseline.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure due to non-ischemic disease (idiopathic cardiomyopathy) or coronary artery disease (CAD) that can not be revascularized.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in the Minnesota Living with Heart Failure Questionnaire. | 6 months

SECONDARY OUTCOMES:
Heart Failure Symptoms | Days 90, 180 and 360
  Heart Failure Symptoms as assessed by New York Heart Association (NYHA) Functional Classification
LVESV/LVEDV | Day 180
  Left ventricular function assessed by contrast Echocardiography
LVEF assessed by contrast Echocardiography | Day 180
  Left ventricular function assessed by contrast Echocardiography
Treadmill exercise test | Day 180
Angina Symptoms | Days 90, 180 and 360
  Angina Symptoms as measured by Canadian Cardiovascular Society Grading System for exertion-induced angina

OTHER OUTCOMES:
MACEs defined as cardiac death, myocardial infarction or hospitalization for heart failure. | Ongoing evaluation from Day 1 through Month 60

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, Study Chair — Cytori Therapeutics